CLINICAL TRIAL: NCT06523231
Title: Safety and Immunogenicity of a Second Generation Shigella Bioconjugate Vaccine: a Phase II Randomized, Controlled, and Blinded Study in 9-month-old Infants
Brief Title: Study to Expand Safety and Immunogenicity Data With Shigella Bioconjugate Vaccine (Shigella4V2) in 9-month-old Infants.
Acronym: S4V02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S4V02
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary | interventions — MenACWY

STUDY DESIGN:
Intervention Model Description: This phase 2 trial is a single center, randomized, controlled, double-blind. Safety and immunogenicity of the vaccine will be evaluated in infants. Subjects will be vaccinated concurrently, with each group randomized to receive 1 of 2 different vaccine doses, or a control vaccine. Participants will be randomized at a ratio of 8:3, to receive the candidate vaccine (low dose : high dose 4:4) or the control vaccine.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose (Experimental): Participants receive 2 low-dose administrations of the investigational product
  Interventions: Biological: Shigella4V2
- high dose (Experimental): Participants receive 2 high-dose administrations of the investigational product
  Interventions: Biological: Shigella4V2
- Control (Other): Participants receive 2 administrations of MenACWY
  Interventions: Biological: MenACWY

INTERVENTIONS:
Biological: Shigella4V2 — Adjuvanted Shigella4V2 administrated at 2 different doses: low and high.
  Arms: high dose; low dose
Biological: MenACWY — Control vaccine
  Arms: Control

SUMMARY:
In this study, the second-generation tetravalent bioconjugate candidate vaccine Shigella4V2 will be tested to confirm data on its safety and immunogenicity in infants and to identify the best dose of Shigella4V2 in 9-month-old infants.

DETAILED DESCRIPTION:
Shigella4V2 is the second generation of a tetravalent bioconjugate vaccine including O-antigen-polysaccharides of the most predominant Shigella serotypes.

During the study, infants will be randomized to receive 1 of 2 different vaccine doses, or a control vaccine.

Participants will receive a 2-dose schedule. Each vaccine dose is formulated with Aluminium adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 9 months (± 1 month) old at the time of the first vaccination.
* Born full-term (i.e., after a gestation period of 37 to less than 42 full weeks).
* Healthy by medical history, laboratory findings and physical examination before entering into the study (Participants with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Seronegative for HIV, hepatitis B and C (as per screening laboratory tests)
* Resident of Siaya County during the whole trial period.
* Previously completed routine primary vaccinations (6,10 and 14 weeks or thereabouts) to the best knowledge of the participant's parent/guardian. This information will be abstracted from the maternal and child health booklet. All the participant's parent/guardian will be requested to carry this booklet whenever they visit the clinic.
* Signed/thumb printed informed consent, in accordance with local practice, provided by participants' parents or guardian who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Demonstrated comprehension (by the parent/guardian) of the protocol procedures through passing a written/verbal comprehension test with a score of 80% or higher (at least 10 out of 12 questions).

Exclusion Criteria:

* Any clinically significant deviation from the normal range in biochemistry or hematological blood tests.
* Suspected or known hypersensitivity (including allergy) to any of the vaccine components or to previous vaccine, or to medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any confirmed or suspected immunosuppressive or immune-deficient condition.
* Systemic administration of corticosteroids (PO/IV/IM): prednisone ≥20 mg/day, or equivalent for more than 14 consecutive days from birth within 90 days prior to informed consent. Inhaled except for doses > 800 mg/day and topical steroids are allowed.
* Administration of antineoplastic or radiotherapy from birth / within 90 days prior to informed consent. Participants may be on chronic or as needed medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition.
* Known exposure to Shigella during lifetime of the study participant
* Concurrently participating in another clinical study, or participation in the preceding month, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Acute illness with or without fever is a temporary exclusion criterium. Positive malaria test is a temporary exclusion criterion.
* History of any malignancy of lymphoproliferative disorder.
* Parent/guardian known to be part of study personnel or being a close family member to the personnel conducting this study.
* Previous history of significant persistent neutropenia, or drug related Neutropenia.
* Weight-for-age Z score less than -3 Standard Deviations (SD).
* History of any chronic or progressive disease (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease) that according to judgment of the investigator could interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine.
* Any medical, social condition, or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation or impairs the parent's/guardian's ability to give informed consent, increases the risk to the potential participant because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 8 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Safety - Solicited Local and Systemic Adverse Events (AEs) | During 7 days following each vaccination
  Safety and tolerability of the candidate vaccine Shigella4V2 as determined by occurrence, severity, and relationship of solicited AEs
Safety - Unsolicited Adverse Events (AEs) | During 28 days following each vaccination
  Safety and tolerability of the candidate vaccine Shigella4V2 as determined by occurrence, severity, and relationship of unsolicited AEs
Safety - Serious Adverse Events (SAEs) | Throughout the study, up to 9 months
  Safety and tolerability of the candidate vaccine Shigella4V2 as determined by occurrence, severity, and relationship of SAEs
Immunology - change in serum immunoglobulin G (IgG) | From first vaccination until 1 month following the second vaccination
  Evaluation of geometric mean titers (GMT) and geometric mean ratios between baseline and 1-month post 2nd vaccination (GMR vs baseline) for serum IgG against the four Shigella serotypes included in the Shigella4V2 bioconjugate.

SECONDARY OUTCOMES:
Safety - clinically significant changes in cell blood count (CBC) with differentials | From first vaccination until 7 days following each vaccination
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in haematological safety parameters
Safety - clinically significant changes in creatinine level | From first vaccination until 7 days following each vaccination
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Safety - clinically significant changes in alanine aminotransferase (ALT) level | From first vaccination until 7 days following each vaccination
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Safety - clinically significant changes in aspartate aminotransferase (AST) level | From first vaccination until 7 days following each vaccination
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Immunogenicity - persistence of serum IgG | From first vaccination until 6 months post 2nd vaccination
  Evaluation of geometric mean titers (GMT) for serum IgG against the four Shigella serotypes included in Shigella4V2 at 6 months post 2nd vaccination.
Immunogenicity - change in serum IgG | From first vaccination until 6 months post 2nd vaccination
  Serum IgG responses and fold-increases between baseline and post-vaccination samples against the four Shigella serotypes included in the Shigella4V2 bioconjugate
Immunogenicity - change in anti-Shigella lipopolysaccharide (LPS) antibody titers | From first vaccination up to 1 month post 2nd vaccination
  Percentage of study participants achieving at least a four-fold increase in anti-Shigella LPS antibody titers (sero-responders) 1-month post 2nd vaccination compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Omore, PhD, Principal Investigator — KEMRI - Center for Global Health Research
Locations (1):
- KEMRI - Center for Global Health Research, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalil IA, Troeger C, Blacker BF, Rao PC, Brown A, Atherly DE, Brewer TG, Engmann CM, Houpt ER, Kang G, Kotloff KL, Levine MM, Luby SP, MacLennan CA, Pan WK, Pavlinac PB, Platts-Mills JA, Qadri F, Riddle MS, Ryan ET, Shoultz DA, Steele AD, Walson JL, Sanders JW, Mokdad AH, Murray CJL, Hay SI, Reiner RC Jr. Morbidity and mortality due to shigella and enterotoxigenic Escherichia coli diarrhoea: the Global Burden of Disease Study 1990-2016. Lancet Infect Dis. 2018 Nov;18(11):1229-1240. doi: 10.1016/S1473-3099(18)30475-4. Epub 2018 Sep 25. PMID 30266330
- [Background] Bengtsson RJ, Simpkin AJ, Pulford CV, Low R, Rasko DA, Rigden DJ, Hall N, Barry EM, Tennant SM, Baker KS. Pathogenomic analyses of Shigella isolates inform factors limiting shigellosis prevention and control across LMICs. Nat Microbiol. 2022 Feb;7(2):251-261. doi: 10.1038/s41564-021-01054-z. Epub 2022 Jan 31. PMID 35102306
- [Background] GBD 2015 LRI Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of lower respiratory tract infections in 195 countries: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Infect Dis. 2017 Nov;17(11):1133-1161. doi: 10.1016/S1473-3099(17)30396-1. Epub 2017 Aug 23. PMID 28843578
- [Background] Luby SP, Rahman M, Arnold BF, Unicomb L, Ashraf S, Winch PJ, Stewart CP, Begum F, Hussain F, Benjamin-Chung J, Leontsini E, Naser AM, Parvez SM, Hubbard AE, Lin A, Nizame FA, Jannat K, Ercumen A, Ram PK, Das KK, Abedin J, Clasen TF, Dewey KG, Fernald LC, Null C, Ahmed T, Colford JM Jr. Effects of water quality, sanitation, handwashing, and nutritional interventions on diarrhoea and child growth in rural Bangladesh: a cluster randomised controlled trial. Lancet Glob Health. 2018 Mar;6(3):e302-e315. doi: 10.1016/S2214-109X(17)30490-4. Epub 2018 Jan 29. PMID 29396217
- [Background] Kotloff KL, Nataro JP, Blackwelder WC, Nasrin D, Farag TH, Panchalingam S, Wu Y, Sow SO, Sur D, Breiman RF, Faruque AS, Zaidi AK, Saha D, Alonso PL, Tamboura B, Sanogo D, Onwuchekwa U, Manna B, Ramamurthy T, Kanungo S, Ochieng JB, Omore R, Oundo JO, Hossain A, Das SK, Ahmed S, Qureshi S, Quadri F, Adegbola RA, Antonio M, Hossain MJ, Akinsola A, Mandomando I, Nhampossa T, Acacio S, Biswas K, O'Reilly CE, Mintz ED, Berkeley LY, Muhsen K, Sommerfelt H, Robins-Browne RM, Levine MM. Burden and aetiology of diarrhoeal disease in infants and young children in developing countries (the Global Enteric Multicenter Study, GEMS): a prospective, case-control study. Lancet. 2013 Jul 20;382(9888):209-22. doi: 10.1016/S0140-6736(13)60844-2. Epub 2013 May 14. PMID 23680352
- [Background] Kotloff KL, Blackwelder WC, Nasrin D, Nataro JP, Farag TH, van Eijk A, Adegbola RA, Alonso PL, Breiman RF, Faruque AS, Saha D, Sow SO, Sur D, Zaidi AK, Biswas K, Panchalingam S, Clemens JD, Cohen D, Glass RI, Mintz ED, Sommerfelt H, Levine MM. The Global Enteric Multicenter Study (GEMS) of diarrheal disease in infants and young children in developing countries: epidemiologic and clinical methods of the case/control study. Clin Infect Dis. 2012 Dec;55 Suppl 4(Suppl 4):S232-45. doi: 10.1093/cid/cis753. PMID 23169936
- [Background] O'Reilly CE, Jaron P, Ochieng B, Nyaguara A, Tate JE, Parsons MB, Bopp CA, Williams KA, Vinje J, Blanton E, Wannemuehler KA, Vulule J, Laserson KF, Breiman RF, Feikin DR, Widdowson MA, Mintz E. Risk factors for death among children less than 5 years old hospitalized with diarrhea in rural western Kenya, 2005-2007: a cohort study. PLoS Med. 2012;9(7):e1001256. doi: 10.1371/journal.pmed.1001256. Epub 2012 Jul 3. PMID 22802736
- [Background] Livio S, Strockbine NA, Panchalingam S, Tennant SM, Barry EM, Marohn ME, Antonio M, Hossain A, Mandomando I, Ochieng JB, Oundo JO, Qureshi S, Ramamurthy T, Tamboura B, Adegbola RA, Hossain MJ, Saha D, Sen S, Faruque AS, Alonso PL, Breiman RF, Zaidi AK, Sur D, Sow SO, Berkeley LY, O'Reilly CE, Mintz ED, Biswas K, Cohen D, Farag TH, Nasrin D, Wu Y, Blackwelder WC, Kotloff KL, Nataro JP, Levine MM. Shigella isolates from the global enteric multicenter study inform vaccine development. Clin Infect Dis. 2014 Oct;59(7):933-41. doi: 10.1093/cid/ciu468. Epub 2014 Jun 23. PMID 24958238
- [Background] Samandari T, Okafor CN. Shigellosis. 2025 Dec 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482337/ PMID 29493962
- [Background] Khan WA, Griffiths JK, Bennish ML. Gastrointestinal and extra-intestinal manifestations of childhood shigellosis in a region where all four species of Shigella are endemic. PLoS One. 2013 May 17;8(5):e64097. doi: 10.1371/journal.pone.0064097. Print 2013. PMID 23691156
- [Background] Shad AA, Shad WA. Shigella sonnei: virulence and antibiotic resistance. Arch Microbiol. 2021 Jan;203(1):45-58. doi: 10.1007/s00203-020-02034-3. Epub 2020 Sep 14. PMID 32929595
- [Background] Puzari M, Sharma M, Chetia P. Emergence of antibiotic resistant Shigella species: A matter of concern. J Infect Public Health. 2018 Jul-Aug;11(4):451-454. doi: 10.1016/j.jiph.2017.09.025. Epub 2017 Oct 20. PMID 29066021
- [Background] Riddle MS, Kaminski RW, Di Paolo C, Porter CK, Gutierrez RL, Clarkson KA, Weerts HE, Duplessis C, Castellano A, Alaimo C, Paolino K, Gormley R, Gambillara Fonck V. Safety and Immunogenicity of a Candidate Bioconjugate Vaccine against Shigella flexneri 2a Administered to Healthy Adults: a Single-Blind, Randomized Phase I Study. Clin Vaccine Immunol. 2016 Dec 5;23(12):908-917. doi: 10.1128/CVI.00224-16. Print 2016 Dec. PMID 27581434
- [Background] Talaat KR, Alaimo C, Martin P, Bourgeois AL, Dreyer AM, Kaminski RW, Porter CK, Chakraborty S, Clarkson KA, Brubaker J, Elwood D, Frolich R, DeNearing B, Weerts H, Feijoo BL, Halpern J, Sack D, Riddle MS, Fonck VG. Human challenge study with a Shigella bioconjugate vaccine: Analyses of clinical efficacy and correlate of protection. EBioMedicine. 2021 Apr;66:103310. doi: 10.1016/j.ebiom.2021.103310. Epub 2021 Apr 13. PMID 33862589
- [Background] Cohen D, Ashkenazi S, Green M, Lerman Y, Slepon R, Robin G, Orr N, Taylor DN, Sadoff JC, Chu C, Shiloach J, Schneerson R, Robbins JB. Safety and immunogenicity of investigational Shigella conjugate vaccines in Israeli volunteers. Infect Immun. 1996 Oct;64(10):4074-7. doi: 10.1128/iai.64.10.4074-4077.1996. PMID 8926071
- [Background] Passwell JH, Ashkenazi S, Banet-Levi Y, Ramon-Saraf R, Farzam N, Lerner-Geva L, Even-Nir H, Yerushalmi B, Chu C, Shiloach J, Robbins JB, Schneerson R; Israeli Shigella Study Group. Age-related efficacy of Shigella O-specific polysaccharide conjugates in 1-4-year-old Israeli children. Vaccine. 2010 Mar 2;28(10):2231-2235. doi: 10.1016/j.vaccine.2009.12.050. Epub 2010 Jan 5. PMID 20056180
- [Background] Ashkenazi S, Passwell JH, Harlev E, Miron D, Dagan R, Farzan N, Ramon R, Majadly F, Bryla DA, Karpas AB, Robbins JB, Schneerson R. Safety and immunogenicity of Shigella sonnei and Shigella flexneri 2a O-specific polysaccharide conjugates in children. J Infect Dis. 1999 Jun;179(6):1565-8. doi: 10.1086/314759. PMID 10228084